CLINICAL TRIAL: NCT02795767
Title: A Multicenter, Open-Label, Phase III Clinical Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of Subcutaneous Administration of Emicizumab in Hemophilia A Pediatric Patients With Inhibitors
Brief Title: A Study of Emicizumab Administered Subcutaneously (SC) in Pediatric Participants With Hemophilia A and Factor VIII (FVIII) Inhibitors
Acronym: HAVEN 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BH29992; 2016-000073-21 (EudraCT Number)
Expanded Access: NCT03154437 (Approved for marketing)
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Results first posted 2019-04-10 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: 1.5 mg/kg Emicizumab QW (Experimental): Participants will receive emicizumab at a loading dose of 3 milligrams per kilogram (mg/kg) QW SC for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg QW SC for a minimum of 52 weeks, or until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria set forth in the protocol, whichever occurs first.
  Interventions: Drug: Emicizumab
- Cohort B: 3 mg/kg Emicizumab Q2W (Experimental): Participants will receive emicizumab at a loading dose of 3 mg/kg QW SC for the first 4 weeks followed by a maintenance dose of 3 mg/kg every 2 weeks (Q2W) SC for a minimum of 52 weeks, or until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria set forth in the protocol, whichever occurs first.
  Interventions: Drug: Emicizumab
- Cohort C: 6 mg/kg Emicizumab Q4W (Experimental): Participants will receive emicizumab at a loading dose of 3 mg/kg QW SC for the first 4 weeks followed by a maintenance dose of 6 mg/kg every 4 weeks (Q4W) SC for a minimum of 52 weeks, or until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria set forth in the protocol, whichever occurs first.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Emicizumab will be administered as per the schedule specified in the respective arm.
  Other Names: Hemlibra; RO5534262; RG6013; ACE910

SUMMARY:
This non-randomized, multicenter, open-label, Phase III clinical study will evaluate the efficacy, safety, and pharmacokinetics of emicizumab administered subcutaneously initially once weekly (QW) in pediatric participants with hemophilia A with FVIII inhibitors. This study will open two additional non-randomized cohorts to investigate once every 2 weeks (Q2W) and once every 4 weeks (Q4W) regimens in pediatric participants.

ELIGIBILITY:
Inclusion Criteria:

* Children less than (<) 12 years of age, with allowance for participants 12 to 17 years of age who weigh <40 kilograms (kg) (Cohort A only); and participants <2 years of age will be allowed to participate only after the protocol-defined interim data review criteria are met (Cohort A only)
* Diagnosis of congenital hemophilia A of any severity and documented history of high-titer inhibitor (that is [i.e.], greater than or equal to [>/=] 5 bethesda units [BU])
* Requires treatment with bypassing agents
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than hemophilia A
* Ongoing (or planning to receive during the study) immune tolerance induction (ITI) therapy or prophylaxis treatment with FVIII
* Previous (in the past 12 months) or current treatment for thromboembolic disease or signs of thromboembolic disease
* Other disease that may increase risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapy or components of the emicizumab injection
* Known infection with human immunodeficiency virus (HIV) or hepatitis B or C virus
* Use of systemic immunomodulators at enrollment or planned use during the study period
* Planned surgery (excluding minor procedures such as tooth extraction or incision and drainage) during the study
* Inability (or unwillingness by caregiver) to receive (allow receipt of) blood or blood products (or any standard-of-care treatment for a life-threatening condition)
* Participants who are at high risk for thrombotic microangiopathy (TMA) (e.g., have a previous medical or family history of TMA), in the investigator's judgement

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- United States (8):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Colorado Denver, Children's Hospital, Aurora, Colorado
  - Children'S Healthcare of Atlanta, Atlanta, Georgia
  - Rush Medical Center, Chicago, Illinois
  - Children's Hospital of Michigan; Pediatrics, Detroit, Michigan
  - North Shore/Long Island Jewish PRIME; Pediatric Hematology/Oncology & Stem Cell Transplantation, New Hyde Park, New York
  - Oregon Health & Science Uni ; Dept of Pediatrics, Portland, Oregon
  - Bloodworks Northwest (formerly Puget Sound Blood Center); Hemophilia, Seattle, Washington
- ICIC, San José, Costa Rica
- France (3):
  - Hopital Cardio-vasculaire Louis Pradel; Hemostase clinique, Bron
  - CH de Bicetre; Centre de Traitement d' Hemophilie, Le Kremlin-Bicêtre
  - Groupe Hospitalier Necker Enfants Malades, Paris
- Universitätsklinikum Bonn; Institut für Experimentelle Hämatologie und Transfusionsmedizin, Bonn, Germany
- IRCCS Ca' Granda Ospedale Maggiore Policlinico; Centro Emofilia e Trombosi "Angelo Bianchi e Bonomi", Milan, Lombardy, Italy
- Japan (5):
  - Nagoya University Hospital, Aichi
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - Nara Medical University Hospital, Nara
  - Shizuoka Children's Hospital, Shizuoka
  - Ogikubo Hospital, Tokyo
- Charlotte Maxeke Johannesburg Hospital; Haemophilia Comprehensive Care Center, Johannesburg, South Africa
- Spain (3):
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
  - Hospital Universitario la Fe; Servicio de Hematologia, Valencia
- Turkey (Türkiye) (4):
  - Adana Acibadem Hospital; Pediatric Hematology, Adana
  - Istanbul Uni Istanbul Medical Faculty, Istanbul
  - Istanbul University, Cerrahpasa Medical Faculty; Pediatrics Department, Istanbul
  - Ege University, School of Medicine; Pediatrics Department, Izmir
- Great Ormond street Hospital for Children NHS Foundation Trust; Haemophilia Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Kruse-Jarres R, Peyvandi F, Oldenburg J, Chang T, Chebon S, Doral MY, Croteau SE, Lambert T, Kempton CL, Pipe SW, Ko RH, Trzaskoma B, Dhalluin C, Bienz NS, Niggli M, Lehle M, Paz-Priel I, Young G, Jimenez-Yuste V. Surgical outcomes in people with hemophilia A taking emicizumab prophylaxis: experience from the HAVEN 1-4 studies. Blood Adv. 2022 Dec 27;6(24):6140-6150. doi: 10.1182/bloodadvances.2022007458. PMID 35939785
- [Derived] Young G, Liesner R, Chang T, Sidonio R, Oldenburg J, Jimenez-Yuste V, Mahlangu J, Kruse-Jarres R, Wang M, Uguen M, Doral MY, Wright LY, Schmitt C, Levy GG, Shima M, Mancuso ME. A multicenter, open-label phase 3 study of emicizumab prophylaxis in children with hemophilia A with inhibitors. Blood. 2019 Dec 12;134(24):2127-2138. doi: 10.1182/blood.2019001869. PMID 31697801

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following completion of accrual to Cohort A: 1.5 mg/kg Emicizumab QW, enrollment was opened to Cohort B: 3 mg/kg Emicizumab Q2W and Cohort C: 6 mg/kg Emicizumab Q4W. Of note, enrollment remained open to Cohort A only for participants who were <2 years old, and enrollment to Cohorts B and C was limited to participants who were 2-11 years old.
Groups:
- Cohort A: 1.5 mg/kg Emicizumab QW: Participants received emicizumab at a loading dose of 3 milligrams per kilogram (mg/kg) once every week (QW) subcutaneously (SC) for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg QW SC for a minimum of 52 weeks, or until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria set forth in the protocol, whichever occurred first.
- Cohort B: 3 mg/kg Emicizumab Q2W: Participants received emicizumab at a loading dose of 3 mg/kg QW subcutaneously (SC) for the first 4 weeks followed by a maintenance dose of 3 mg/kg once every 2 weeks (Q2W) SC for a minimum of 52 weeks, or until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria set forth in the protocol, whichever occurred first.
- Cohort C: 6 mg/kg Emicizumab Q4W: Participants received emicizumab at a loading dose of 3 mg/kg QW subcutaneously (SC) for the first 4 weeks followed by a maintenance dose of 6 mg/kg once every 4 weeks (Q4W) SC for a minimum of 52 weeks, or until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria set forth in the protocol, whichever occurred first.
Period: Overall Study
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Started | 68 | 10 | 10
Received at Least One Dose of Emicizumab | 68 | 10 | 10
Dose Up-Titrated to 3 mg/kg QW | 0 | 0 | 3
Completed 52 Weeks in Study | 67 | 10 | 9
Completed | 67 | 10 | 10
Not Completed | 1 | 0 | 0
Not completed — Received Commercial Emicizumab | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W | Total
Number analyzed (Participants) | 68 | 10 | 10 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (3.6) | 6.9 (3.2) | 7.9 (3.0) | 6.5 (3.5)
Age, Customized [Count of Participants; unit: Participants]
  0 to <2 Years Old | 8 | 0 | 0 | 8
  2 to <6 Years Old | 19 | 3 | 2 | 24
  6 to <12 Years Old | 38 | 7 | 8 | 53
  ≥12 Years Old | 3 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 68 | 10 | 10 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 1 | 7
  Not Hispanic or Latino | 61 | 9 | 9 | 79
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 1 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 11 | 1 | 0 | 12
  White | 39 | 7 | 8 | 54
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 6 | 1 | 0 | 7
Number of Participants with 0, 1, or >1 Target Joint in the Last 24 Weeks Prior to Study Entry [Count of Participants; unit: Participants] — A target joint was defined as a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry.
  Participants
    0 Target Joints | 44 | 3 | 7 | 54
    1 Target Joint | 9 | 6 | 1 | 16
    >1 Target Joint | 15 | 1 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Model-Based Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants <12 Years of Age
Description: The number of treated bleeds over the efficacy period is presented here as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and the first treatment thereafter and before a new bleed starts, are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: From Baseline to 52 weeks; At the primary completion date, the median (min-max) duration of the efficacy period in Cohort A was 57.57 (17.9-92.6) weeks.
Population: All treated participants in Cohort A who were on the same dose of emicizumab for at least 12 weeks and were <12 years of age
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated bleed rate per year | 0.3 [0.17 to 0.50]

2. Primary Outcome: Cohort A: Model-Based Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants <12 Years of Age
Description: The number of all bleeds over the efficacy period is presented here as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in followup times (i.e., the time that each participant stays in the study). In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
all bleed rate per year | 3.2 [1.94 to 5.22]

3. Primary Outcome: Cohort A: Model-Based Annualized Bleed Rate (ABR) for Treated Spontaneous Bleeds in Treated Participants <12 Years of Age
Description: The number of treated spontaneous bleeds over the efficacy period is presented here as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A bleed is classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "treated spontaneous bleed" is a spontaneous bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Treated bleeds that fulfilled the 72-hour rule were included in the analysis of spontaneous bleeds. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: treated spontaneous bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated spontaneous bleed rate per year | 0.0 [0.0 to 0.1]

4. Primary Outcome: Cohort A: Model-Based Annualized Bleed Rate (ABR) for Treated Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of treated joint bleeds over the efficacy period is presented here as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A "joint bleed" is defined as a bleed with type reported as "joint" and with at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline. A "treated joint bleed" is a joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Only treated bleeds that fulfilled the 72-hour rule were included in the analysis of treated joint bleeds, excluding bleeds due to surgery/procedure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: treated joint bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated joint bleed rate per year | 0.2 [0.08 to 0.29]

5. Primary Outcome: Cohort A: Model-Based Annualized Bleed Rate (ABR) for Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of treated target joint bleeds over the efficacy period is presented here as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A "target joint bleed" is defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry. A "treated target joint bleed" is a target joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: treated target joint bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated target joint bleed rate per year | NA [NA to NA] — The model-based ABR and 95% CI were not estimable because too few events had occurred over the efficacy period to calculate values using the negative binomial regression model; 95.4% of participants in this cohort had 0 treated target joint bleeds.

6. Primary Outcome: Cohort A: Mean Calculated Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants <12 Years of Age
Description: The number of treated bleeds over the efficacy period is presented here as a calculated ABR that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and the first treatment thereafter and before a new bleed starts, are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: treated bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated bleed rate per year | 0.3 [0.00 to 4.31]

7. Primary Outcome: Cohort A: Mean Calculated Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants <12 Years of Age
Description: The number of all bleeds over the efficacy period is presented here as a calculated ABR that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
all bleed rate per year | 3.2 [0.70 to 9.04]

8. Primary Outcome: Cohort A: Mean Calculated Annualized Bleed Rate (ABR) for Treated Spontaneous Bleeds in Treated Participants <12 Years of Age
Description: The number of treated spontaneous bleeds over the efficacy period is presented here as a calculated ABR that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A bleed is classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "treated spontaneous bleed" is a spontaneous bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Treated bleeds that fulfilled the 72-hour rule were included in the analysis of spontaneous bleeds. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: treated spontaneous bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated spontaneous bleed rate per year | 0.0 [0.00 to 3.74]

9. Primary Outcome: Cohort A: Mean Calculated Annualized Bleed Rate (ABR) for Treated Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of treated joint bleeds over the efficacy period is presented here as a calculated ABR that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A "joint bleed" is defined as a bleed with type reported as "joint" and with at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline. A "treated joint bleed" is a joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Only treated bleeds that fulfilled the 72-hour rule were included in the analysis of treated joint bleeds, excluding bleeds due to surgery/procedure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: treated joint bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated joint bleed rate per year | 0.2 [0.00 to 4.01]

10. Primary Outcome: Cohort A: Mean Calculated Annualized Bleed Rate (ABR) for Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of treated target joint bleeds over the efficacy period is presented here as a calculated ABR that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A "target joint bleed" is defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry. A "treated target joint bleed" is a target joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: treated target joint bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated target joint bleed rate per year | 0.1 [0.00 to 3.84]

11. Primary Outcome: Cohort A: Median Calculated Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: treated bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated bleed rate per year | 0.0 [0.00 to 0.00]

12. Primary Outcome: Cohort A: Median Calculated Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 7
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: all bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
all bleed rate per year | 0.6 [0.00 to 2.92]

13. Primary Outcome: Cohort A: Median Calculated Annualized Bleed Rate (ABR) for Treated Spontaneous Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: treated spontaneous bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated spontaneous bleed rate per year | 0.0 [0.00 to 0.00]

14. Primary Outcome: Cohort A: Median Calculated Annualized Bleed Rate (ABR) for Treated Joint Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 9
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: treated joint bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated joint bleed rate per year | 0.0 [0.00 to 0.00]

15. Primary Outcome: Cohort A: Median Calculated Annualized Bleed Rate (ABR) for Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 10
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: treated target joint bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
treated target joint bleed rate per year | 0.0 [0.00 to 0.00]

16. Primary Outcome: Cohort A: Percentage of Participants by Categorized Number of Treated Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: The percentage of participants by categorized number of treated bleeds over the efficacy period is presented here. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and the first treatment thereafter and before a new bleed starts, are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
percentage of participants
  0 Bleeds | 76.9 [64.8 to 86.5]
  0-3 Bleeds | 100.0 [94.5 to 100.0]
  0-10 Bleeds | 100.0 [94.5 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 5.5]

17. Primary Outcome: Cohort A: Percentage of Participants by Categorized Number of All Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: The percentage of participants by categorized number of all bleeds over the efficacy period is presented here. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
percentage of participants
  0 Bleeds | 49.2 [36.6 to 61.9]
  0-3 Bleeds | 72.3 [59.8 to 82.7]
  0-10 Bleeds | 92.3 [83.0 to 97.5]
  >10 Bleeds | 7.7 [2.5 to 17.0]

18. Primary Outcome: Cohort A: Percentage of Participants by Categorized Number of Treated Spontaneous Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: The percentage of participants by categorized number of treated spontaneous bleeds over the efficacy period is presented here. A bleed is classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "treated spontaneous bleed" is a spontaneous bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Treated bleeds that fulfilled the 72-hour rule were included in the analysis of spontaneous bleeds. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
percentage of participants
  0 Bleeds | 96.9 [89.3 to 99.6]
  0-3 Bleeds | 100.0 [94.5 to 100.0]
  0-10 Bleeds | 100.0 [94.5 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 5.5]

19. Primary Outcome: Cohort A: Percentage of Participants by Categorized Number of Treated Joint Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: The percentage of participants by categorized number of treated joint bleeds over the efficacy period is presented here. A "joint bleed" is defined as a bleed with type reported as "joint" and with at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline. A "treated joint bleed" is a joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Only treated bleeds that fulfilled the 72-hour rule were included in the analysis of treated joint bleeds, excluding bleeds due to surgery/procedure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
percentage of participants
  0 Bleeds | 84.6 [73.5 to 92.4]
  0-3 Bleeds | 100.0 [94.5 to 100.0]
  0-10 Bleeds | 100.0 [94.5 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 5.5]

20. Primary Outcome: Cohort A: Percentage of Participants by Categorized Number of Treated Target Joint Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: The percentage of participants by categorized number of treated target joint bleeds over the efficacy period is presented here. A "target joint bleed" is defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry. A "treated target joint bleed" is a target joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 65
percentage of participants
  0 Bleeds | 95.4 [87.1 to 99.0]
  0-3 Bleeds | 100.0 [94.5 to 100.0]
  0-10 Bleeds | 100.0 [94.5 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 5.5]

21. Secondary Outcome: Cohorts B and C: Model-Based Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants <12 Years of Age
Description: The number of treated bleeds over the efficacy period is presented as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and the first treatment thereafter and before a new bleed starts, are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: From Baseline to 24 weeks; At the primary completion date, the median (min-max) duration of the efficacy periods in Cohorts B and C were 21.29 (18.6-24.1) weeks and 19.86 (8.9-24.1) weeks, respectively.
Population: All treated participants in Cohorts B and C who were on the same dose of emicizumab for at least 12 weeks and were <12 years of age
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated bleed rate per year | 0.2 [0.03 to 1.72] | 2.2 [0.69 to 6.81]

22. Secondary Outcome: Cohorts B and C: Model-Based Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants <12 Years of Age
Description: The number of all bleeds over the efficacy period is presented as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
all bleed rate per year | 1.5 [0.62 to 3.40] | 3.8 [1.42 to 10.11]

23. Secondary Outcome: Cohorts B and C: Model-Based Annualized Bleed Rate (ABR) for Treated Spontaneous Bleeds in Treated Participants <12 Years of Age
Description: The number of treated spontaneous bleeds over the efficacy period is presented as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A bleed is classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "treated spontaneous bleed" is a spontaneous bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Treated bleeds that fulfilled the 72-hour rule were included in the analysis of spontaneous bleeds. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: treated spontaneous bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated spontaneous bleed rate per year | NA [NA to NA] — The model-based ABR and 95% CI were not estimable because too few events had occurred over the efficacy period to calculate values using the negative binomial regression model; 100% of participants in this cohort had 0 treated spontaneous bleeds. | 0.8 [0.05 to 12.00]

24. Secondary Outcome: Cohorts B and C: Model-Based Annualized Bleed Rate (ABR) for Treated Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of treated joint bleeds over the efficacy period is presented as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A "joint bleed" is defined as a bleed with type reported as "joint" and with at least one of the following symptoms: increasing swelling or warmth of the skin over the joint and/or increasing pain, decreased range of motion, or difficulty using the joint compared with baseline. A "treated joint bleed" is a joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Only treated bleeds that fulfilled the 72-hour rule were included in the analysis of treated joint bleeds, excluding bleeds due to surgery/procedure.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: treated joint bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated joint bleed rate per year | 0.2 [0.03 to 1.72] | 1.7 [0.60 to 4.89]

25. Secondary Outcome: Cohorts B and C: Model-Based Annualized Bleed Rate (ABR) for Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of treated target joint bleeds over the efficacy period is presented as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times (i.e., the time that each participant stays in the study). A "target joint bleed" is defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry. A "treated target joint bleed" is a target joint bleed that also fulfills the conditions of a treated bleed (see ABR for Treated Bleeds for the definition). Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: treated target joint bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated target joint bleed rate per year | 0.2 [0.03 to 1.72] | 0.5 [0.05 to 5.88]

26. Secondary Outcome: Cohorts B and C: Mean Calculated Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 6
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: treated bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated bleed rate per year | 0.2 [0.00 to 4.13] | 2.5 [0.43 to 8.06]

27. Secondary Outcome: Cohorts B and C: Mean Calculated Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 7
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
all bleed rate per year | 1.5 [0.10 to 6.36] | 4.0 [1.09 to 10.25]

28. Secondary Outcome: Cohorts B and C: Mean Calculated Annualized Bleed Rate (ABR) for Treated Spontaneous Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 8
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: treated spontaneous bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated spontaneous bleed rate per year | 0.0 [NA to 3.69] — The lower limit of the 95% CI could not be estimated because too few events had occurred over the efficacy period to calculate it; 100% of participants in this cohort had 0 treated spontaneous bleeds. | 0.8 [0.01 to 5.20]

29. Secondary Outcome: Cohorts B and C: Mean Calculated Annualized Bleed Rate (ABR) for Treated Joint Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 9
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: treated joint bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated joint bleed rate per year | 0.2 [0.00 to 4.13] | 1.9 [0.23 to 7.14]

30. Secondary Outcome: Cohorts B and C: Mean Calculated Annualized Bleed Rate (ABR) for Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 10
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (95% Confidence Interval); unit: treated target joint bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated target joint bleed rate per year | 0.2 [0.00 to 4.13] | 0.5 [0.00 to 4.72]

31. Secondary Outcome: Cohorts B and C: Median Calculated Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 6
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: treated bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated bleed rate per year | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 3.26]

32. Secondary Outcome: Cohorts B and C: Median Calculated Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 7
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: all bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
all bleed rate per year | 0.0 [0.00 to 2.81] | 1.6 [0.00 to 4.84]

33. Secondary Outcome: Cohorts B and C: Median Calculated Annualized Bleed Rate (ABR) for Treated Spontaneous Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 8
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: treated spontaneous bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated spontaneous bleed rate per year | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]

34. Secondary Outcome: Cohorts B and C: Median Calculated Annualized Bleed Rate (ABR) for Treated Joint Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 9
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: treated joint bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated joint bleed rate per year | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 3.26]

35. Secondary Outcome: Cohorts B and C: Median Calculated Annualized Bleed Rate (ABR) for Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 10
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: treated target joint bleed rate per year
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
treated target joint bleed rate per year | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]

36. Secondary Outcome: Cohorts B and C: Percentage of Participants by Categorized Number of Treated Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: as for outcome 16
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
percentage of participants
  0 Bleeds | 90.0 [55.5 to 99.7] | 60.0 [26.2 to 87.8]
  0-3 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  0-10 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

37. Secondary Outcome: Cohorts B and C: Percentage of Participants by Categorized Number of All Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: as for outcome 17
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
percentage of participants
  0 Bleeds | 60.0 [26.2 to 87.8] | 50.0 [18.7 to 81.3]
  0-3 Bleeds | 100.0 [69.2 to 100.0] | 90.0 [55.5 to 99.7]
  0-10 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

38. Secondary Outcome: Cohorts B and C: Percentage of Participants by Categorized Number of Treated Spontaneous Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: as for outcome 18
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
percentage of participants
  0 Bleeds | 100.0 [69.2 to 100.0] | 90.0 [55.5 to 99.7]
  0-3 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  0-10 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

39. Secondary Outcome: Cohorts B and C: Percentage of Participants by Categorized Number of Treated Joint Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: as for outcome 19
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
percentage of participants
  0 Bleeds | 90.0 [55.5 to 99.7] | 60.0 [26.2 to 87.8]
  0-3 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  0-10 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

40. Secondary Outcome: Cohorts B and C: Percentage of Participants by Categorized Number of Treated Target Joint Bleeds Over the Efficacy Period in Treated Participants <12 Years of Age
Description: as for outcome 20
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 10 | 10
percentage of participants
  0 Bleeds | 90.0 [55.5 to 99.7] | 90.0 [55.5 to 99.7]
  0-3 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  0-10 Bleeds | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0]
  >10 Bleeds | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

41. Secondary Outcome: Cohort A: Intra-Participant Comparison of the Model-Based ABR for Treated Bleeds on Study Versus Pre-Study in Treated Participants <12 Years of Age From the Non-Interventional Study (NIS) Population
Description: This is an intra-participant comparison of the model-based annualized bleeding rate (ABR) for treated bleeds (i.e., number of treated bleeds over efficacy period using negative binomial regression model) on study versus pre-study in the NIS population who had previously participated in study BH29768 (NCT02476942). A "treated bleed" is a bleed directly followed by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and first treatment thereafter are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: Up to 24 weeks in NIS BH29768 (NCT02476942) prior to study entry and from Baseline to 52 weeks on this study; At primary completion date, the median (min-max) duration of the efficacy period in the NIS population was 88.57 (55.9-92.6) weeks.
Population: Treated participants <12 years of age who had participated in NIS BH29768 (NCT02476942) prior to enrollment in this study and were on the same dose of emicizumab for at least 12 weeks in this study
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Groups:
- Cohort A NIS Population (<12 Years): Bypassing Agents: This group includes historical data from participants <12 years old who had participated in the non-interventional study (NIS) BH29768 (NCT02476942) in which they had received prophylactic or episodic treatment with bypassing agents and had been followed for a minimum of 24 weeks on the NIS prior to enrollment in Cohort A of this study (BH29992).
- Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW: Participants <12 years old who had previously received prophylactic or episodic treatment with bypassing agents in NIS BH29768 (NCT02476942) and were enrolled in Cohort A of this study (BH29992) received emicizumab at a loading dose of 3 milligrams per kilogram (mg/kg) once every week (QW) subcutaneously (SC) for the first 4 weeks followed by a maintenance dose of 1.5 mg/kg emicizumab QW SC for a minimum of 52 weeks, or until unacceptable toxicity, discontinuation from the study due to any cause, or other criteria set forth in the protocol, whichever occurred first.
Arm/Group | Cohort A NIS Population (<12 Years): Bypassing Agents | Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 18 | 18
treated bleed rate per year | 19.9 [15.33 to 25.85] | 0.2 [0.11 to 0.49]
Statistical Analysis 1: Comparison: Cohort A NIS Population (<12 Years): Bypassing Agents vs Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW; Test type: Other; ABR Ratio = 0.01, 95% CI 2-sided [0.006 to 0.023] — Emicizumab QW is the numerator and Prophylactic/Episodic Bypassing Agent is the denominator

42. Secondary Outcome: Cohort A: Intra-Participant Comparison of the Model-Based ABR for All Bleeds on Study Versus Pre-Study in Treated Participants <12 Years of Age From the NIS Population
Description: This is an intra-participant comparison of the model-based annualized bleeding rate (ABR) for all bleeds (i.e., number of all bleeds over efficacy period using negative binomial regression model) on study versus pre-study in the NIS population who had previously participated in study BH29768 (NCT02476942). In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Cohort A NIS Population (<12 Years): Bypassing Agents | Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 18 | 18
all bleed rate per year | 31.9 [22.68 to 44.81] | 3.3 [1.45 to 7.53]
Statistical Analysis 1: Comparison: Cohort A NIS Population (<12 Years): Bypassing Agents vs Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW; Test type: Other; ABR Ratio = 0.10, 95% CI 2-sided [0.051 to 0.210] — Emicizumab QW is the numerator and Prophylactic/Episodic Bypassing Agent is the denominator

43. Secondary Outcome: Cohort A: Intra-Participant Comparison of the Median Calculated ABR for Treated Bleeds on Study Versus Pre-Study in Treated Participants <12 Years of Age From the NIS Population
Description: This is an intra-participant comparison of the calculated ABR for treated bleeds (annualized per participant using the following formula: ABR = [number of bleeds/number of days during the efficacy period] x 365.25) on study versus pre-study in the NIS population who had previously participated in study BH29768 (NCT02476942). A "treated bleed" is a bleed directly followed by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and first treatment thereafter are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: treated bleed rate per year
Arm/Group | Cohort A NIS Population (<12 Years): Bypassing Agents | Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 18 | 18
treated bleed rate per year | 16.2 [11.49 to 25.78] | 0.0 [0.00 to 0.56]

44. Secondary Outcome: Cohort A: Intra-Participant Comparison of the Median Calculated ABR for All Bleeds on Study Versus Pre-Study in Treated Participants <12 Years of Age From the NIS Population
Description: This is an intra-participant comparison of the calculated annualized bleeding rate (ABR) for all bleeds (annualized for each participant using the following formula: ABR = [number of bleeds/number of days during the efficacy period] x 365.25) on study versus pre-study in the NIS population who had previously participated in study BH29768 (NCT02476942). In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: all bleed rate per year
Arm/Group | Cohort A NIS Population (<12 Years): Bypassing Agents | Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 18 | 18
all bleed rate per year | 21.3 [14.18 to 44.47] | 1.1 [0.00 to 2.30]

45. Secondary Outcome: Cohort A: Intra-Participant Comparison of Percentage of Participants by Categorized Number of Treated Bleeds on Study Versus Pre-Study in Treated Participants <12 Years of Age From the NIS Population
Description: This is an intra-participant comparison of the percentage of participants by categorized number of treated bleeds over the efficacy period on study versus pre-study in the NIS population who had previously participated in study BH29768 (NCT02476942). A "treated bleed" is a bleed directly followed by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and first treatment thereafter are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A NIS Population (<12 Years): Bypassing Agents | Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 18 | 18
percentage of participants
  0 Bleeds | 5.6 [0.1 to 27.3] | 72.2 [46.5 to 90.3]
  0-3 Bleeds | 16.7 [3.6 to 41.4] | 100.0 [81.5 to 100.0]
  0-10 Bleeds | 66.7 [41.0 to 86.7] | 100.0 [81.5 to 100.0]
  >10 Bleeds | 33.3 [13.3 to 59.0] | 0.0 [0.0 to 18.5]

46. Secondary Outcome: Cohort A: Intra-Participant Comparison of Percentage of Participants by Categorized Number of All Bleeds on Study Versus Pre-Study in Treated Participants <12 Years of Age From the NIS Population
Description: This is an intra-participant comparison of the percentage of participants by categorized number of all bleeds over the efficacy period on study versus pre-study in the NIS population who had previously participated in study BH29768 (NCT02476942). In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: as for outcome 41
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A NIS Population (<12 Years): Bypassing Agents | Cohort A NIS Population (<12 Years): 1.5 mg/kg Emicizumab QW
Number analyzed (Participants) | 18 | 18
percentage of participants
  0 Bleeds | 0.0 [0.0 to 18.5] | 33.3 [13.3 to 59.0]
  0-3 Bleeds | 11.1 [1.4 to 34.7] | 72.2 [46.5 to 90.3]
  0-10 Bleeds | 44.4 [21.5 to 69.2] | 83.3 [58.6 to 96.4]
  >10 Bleeds | 55.6 [30.8 to 78.5] | 16.7 [3.6 to 41.4]

47. Secondary Outcome: Model-Based Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants ≥12 Years of Age and <40 kg Body Weight
Description: as for outcome 1
Time Frame: From Baseline to 52 weeks
Population: All participants who received at least one dose of emicizumab and were ≥12 years old and weighed <40 kg at the time of informed consent; none of the participants enrolled in Cohorts B and C fit these criteria.
Measure: Number (95% Confidence Interval); unit: treated bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 3 | 0 | 0
treated bleed rate per year | 0.8 [0.25 to 2.40] |  |

48. Secondary Outcome: Model-Based Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants ≥12 Years of Age and <40 kg Body Weight
Description: The number of all bleeds over the efficacy period is presented as a model-based ABR that was analyzed using a negative binomial regression model with efficacy period as an offset to account for the difference in followup times (i.e., the time that each participant stays in the study). In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: From Baseline to 52 weeks
Population: as for outcome 47
Measure: Number (95% Confidence Interval); unit: all bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 3 | 0 | 0
all bleed rate per year | 1.4 [0.49 to 4.16] |  |

49. Secondary Outcome: Median Calculated Annualized Bleed Rate (ABR) for Treated Bleeds in Treated Participants ≥12 Years of Age and <40 kg Body Weight
Description: as for outcome 6
Time Frame: From Baseline to 52 weeks
Population: as for outcome 47
Measure: Median (Inter-Quartile Range); unit: treated bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 3 | 0 | 0
treated bleed rate per year | 0.9 [0.00 to 1.14] |  |

50. Secondary Outcome: Median Calculated Annualized Bleed Rate (ABR) for All Bleeds in Treated Participants ≥12 Years of Age and <40 kg Body Weight
Description: as for outcome 7
Time Frame: From Baseline to 52 weeks
Population: as for outcome 47
Measure: Median (Inter-Quartile Range); unit: all bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 3 | 0 | 0
all bleed rate per year | 0.9 [0.00 to 2.84] |  |

51. Secondary Outcome: Number of Treated Bleeds Over Time in Participants With Dose Up-Titration
Description: The number of treated bleeds over time was to be analyzed in participants whose emicizumab maintenance dose was up-titrated to 3 mg/kg QW if they had experienced suboptimal bleeding control on emicizumab at steady-state, per protocol criteria. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. A bleed and the first treatment thereafter and before a new bleed starts, are considered to be pairs, with the following exception: if multiple bleeds occur on the same calendar day, the subsequent treatment is considered to apply for each of these multiple bleeds. The 72-hour rule was implemented: two bleeds of the same type and at the same anatomical location are counted as one bleed if the second bleed occurs within 72 hours from the last treatment for the first bleed. Bleeds due to surgery/procedure are excluded.
Time Frame: From Baseline to study completion (up to at least 52 weeks)
Population: All participants with emicizumab dose up-titration; At study completion, 0 participants in Cohorts A and B and 3 participants in Cohort C had their emicizumab dose up-titrated over the course of this clinical trial. Data were not aggregated for this outcome measure because it was not part of the pre-specified analysis plan and because of the limited sample size. The results will not be disclosed on an individual patient level because of data privacy concerns.
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 0 | 0 | 0

52. Secondary Outcome: Number of All Bleeds Over Time in Participants With Dose Up-Titration
Description: The number of all bleeds over time was to be analyzed in participants whose emicizumab maintenance dose was up-titrated to 3 mg/kg QW if they had experienced suboptimal bleeding control on emicizumab at steady-state, per protocol criteria. In this outcome measure, all bleeds are included, irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. As "all bleeds" comprises both treated and non-treated bleeds, the 72-hour rule was implemented separately for treated and non-treated bleeds. For treated bleeds, the 72-hour rule was implemented exactly as defined for the "treated bleeds" outcome measure. For non-treated bleeds, the 72-hour rule was implemented by calculating a treatment-free period of 72 hours from the bleed itself.
Time Frame: From Baseline to study completion (up to at least 52 weeks)
Population: as for outcome 51
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 0 | 0 | 0

53. Secondary Outcome: Long-Term Efficacy of Emicizumab in All Cohorts: Model-Based Annualized Bleed Rate (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of bleeds over the efficacy period was shown as a model-based ABR that used a negative binomial regression model with efficacy period as an offset to account for the difference in follow-up times. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. "All bleeds" included bleeds irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. Bleeds are classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "joint bleed" is defined as a bleed occurring in a joint. A "target joint bleed" is defined as a joint bleed in a target joint (≥3 bleeds have occurred over the last 24 weeks prior to study entry).
Time Frame: From Baseline to study completion (median [min-max] duration of the efficacy periods in Cohorts A, B, and C were 92.29 [36.1-187.7] weeks, 68.21 [56.7-129.4] weeks, and 69.43 [8.9-144.3] weeks, respectively)
Population: All treated participants in Cohorts A, B, and C who were on the same dose of emicizumab for at least 12 weeks and were <12 years of age
Measure: Number (95% Confidence Interval); unit: bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 65 | 10 | 10
bleed rate per year
  Treated Bleeds | 0.3 [0.19 to 0.43] | 0.2 [0.06 to 0.54] | 1.8 [0.32 to 10.59]
  All Bleeds | 3.0 [1.93 to 4.55] | 0.8 [0.42 to 1.54] | 2.4 [0.78 to 7.51]
  Treated Spontaneous Bleeds | 0.01 [0.01 to 0.07] | NA [NA to NA] — The model-based ABR and 95% CI were not estimable because too few events had occurred over the efficacy period to calculate values using the negative binomial regression model; 100% of participants in this cohort had 0 treated spontaneous bleeds. | 0.9 [0.08 to 9.93]
  Treated Joint Bleeds | 0.2 [0.09 to 0.25] | 0.2 [0.06 to 0.54] | 1.3 [0.25 to 7.11]
  Treated Target Joint Bleeds | 0.1 [0.01 to 0.30] | 0.1 [0.03 to 0.47] | 0.5 [0.02 to 13.77]

54. Secondary Outcome: Long-Term Efficacy of Emicizumab in All Cohorts: Mean Calculated Annualized Bleed Rate (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: The number of treated bleeds over the efficacy period is presented here as a calculated ABR that was annualized for each participant using the following formula: ABR = (number of bleeds/number of days during the efficacy period) x 365.25. A bleed is considered a "treated bleed" if it is directly followed (i.e., no intervening bleed) by a hemophilia medication reported to be a "treatment for bleed", irrespective of time between treatment and the preceding bleed. "All bleeds" included bleeds irrespective of treatment with coagulation factors, with the following exception: bleeds due to surgery/procedure are excluded. Bleeds are classified as "spontaneous" if there is no other known contributing factor such as trauma or procedure/surgery. A "joint bleed" is defined as a bleed with type reported as "joint". A "target joint bleed" is defined as a joint bleed in a target joint, which is a joint location where at least 3 bleeds have occurred over the last 24 weeks prior to study entry.
Time Frame: as for outcome 53
Population: as for outcome 53
Measure: Mean (95% Confidence Interval); unit: bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 65 | 10 | 10
bleed rate per year
  Treated Bleeds | 0.3 [0.00 to 4.25] | 0.2 [0.00 to 4.02] | 2.2 [0.32 to 7.59]
  All Bleeds | 3.0 [0.61 to 8.74] | 0.8 [0.01 to 5.17] | 3.0 [0.63 to 8.82]
  Treated Spontaneous Bleeds | 0.0 [0.00 to 3.72] | 0.0 [NA to 3.69] — The lower limit of the 95% CI could not be estimated because too few events had occurred over the efficacy period to calculate it; 100% of participants in this cohort had 0 treated spontaneous bleeds. | 1.0 [0.02 to 5.53]
  Treated Joint Bleeds | 0.1 [0.00 to 3.99] | 0.2 [0.00 to 4.02] | 1.6 [0.14 to 6.65]
  Treated Target Joint Bleeds | 0.1 [0.00 to 3.82] | 0.1 [0.00 to 3.86] | 0.5 [0.00 to 4.65]

55. Secondary Outcome: Long-Term Efficacy of Emicizumab in All Cohorts: Median Calculated Annualized Bleed Rate (ABR) for Treated Bleeds, All Bleeds, Treated Spontaneous Bleeds, Treated Joint Bleeds, and Treated Target Joint Bleeds in Treated Participants <12 Years of Age
Description: as for outcome 54
Time Frame: as for outcome 53
Population: as for outcome 53
Measure: Median (Inter-Quartile Range); unit: bleed rate per year
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 65 | 10 | 10
bleed rate per year
  Treated Bleeds | 0.0 [0.00 to 0.51] | 0.0 [0.00 to 0.40] | 0.0 [0.00 to 3.26]
  All Bleeds | 0.7 [0.00 to 3.11] | 0.8 [0.00 to 0.85] | 0.6 [0.00 to 3.26]
  Treated Spontaneous Bleeds | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Treated Joint Bleeds | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.40] | 0.0 [0.00 to 3.26]
  Treated Target Joint Bleeds | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]

56. Secondary Outcome: Change From Baseline Over Time in the Hemophilia-Specific Quality of Life Short Form (Haemo-QoL-SF) Questionnaire Total Score, as Completed by Treated Participants ≥8 to <12 Years of Age
Description: The Haemo-QoL-SF is a self-reported questionnaire for children ≥8 years of age. It contains 35 items, which cover nine domains considered relevant for the children's health-related quality of life: Physical Health, Feelings, View of Yourself, Family, Friends, Other People, Sports and School, Dealing with Hemophilia, and Treatment. Items are rated with five respective response options: never, seldom, sometimes, often, and always. The Total Score is derived from the scores for all domains and ranges from 0 to 100, with a lower score reflective of better health-related quality of life.
Time Frame: Baseline (Week 1), Weeks 13, 25, 37, 49, 57, 81, 105, 129, 153, and 177, and at study completion [SC] or early discontinuation [ED] (up to 188 weeks)
Population: All treated participants ≥8 to <12 years of age; at each timepoint, the number analyzed is the number of participants who completed a sufficient number of questionnaire items.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 22 | 6 | 6
score on a scale
  Baseline (value at visit): number analyzed (Participants) | 18 | 6 | 6
  Baseline (value at visit) | 33.37 [25.15 to 41.60] | 25.60 [18.29 to 32.90] | 25.12 [9.85 to 40.39]
  Change from Baseline at Week 13: number analyzed (Participants) | 18 | 6 | 5
  Change from Baseline at Week 13 | -7.02 [-12.08 to -1.96] | -9.17 [-15.59 to -2.75] | 0.29 [-23.12 to 23.69]
  Change from Baseline at Week 25: number analyzed (Participants) | 18 | 6 | 4
  Change from Baseline at Week 25 | -9.17 [-15.97 to -2.37] | -13.21 [-23.43 to -2.99] | -14.64 [-42.98 to 13.70]
  Change from Baseline at Week 37: number analyzed (Participants) | 17 | 6 | 3
  Change from Baseline at Week 37 | -11.64 [-16.11 to -7.17] | -15.48 [-24.58 to -6.37] | -17.86 [-71.56 to 35.85]
  Change from Baseline at Week 49: number analyzed (Participants) | 17 | 5 | 3
  Change from Baseline at Week 49 | -9.62 [-13.59 to -5.65] | -15.14 [-25.05 to -5.24] | -16.43 [-67.33 to 34.47]
  Change from Baseline at Week 57: number analyzed (Participants) | 12 | 4 | 2
  Change from Baseline at Week 57 | -11.13 [-17.92 to -4.34] | -16.43 [-25.85 to -7.01] | -25.00 [-215.59 to 165.59]
  Change from Baseline at Week 81: number analyzed (Participants) | 12 | 3 | 0
  Change from Baseline at Week 81 | -11.79 [-20.23 to -3.34] | -14.52 [-31.76 to 2.71] |
  Change from Baseline at Week 105: number analyzed (Participants) | 9 | 3 | 0
  Change from Baseline at Week 105 | -18.57 [-35.25 to -1.90] | -14.76 [-30.76 to 1.24] |
  Change from Baseline at Week 129: number analyzed (Participants) | 7 | 0 | 0
  Change from Baseline at Week 129 | -14.90 [-29.47 to -0.32] |  |
  Change from Baseline at Week 153: number analyzed (Participants) | 4 | 0 | 0
  Change from Baseline at Week 153 | -14.46 [-32.37 to 3.44] |  |
  Change from Baseline at Week 177: number analyzed (Participants) | 2 | 0 | 0
  Change from Baseline at Week 177 | -5.36 [-118.81 to 108.09] |  |
  Change from Baseline at SC or ED: number analyzed (Participants) | 11 | 3 | 2
  Change from Baseline at SC or ED | -13.05 [-22.31 to -3.79] | -21.43 [-37.40 to -5.46] | -28.21 [-241.50 to 185.07]

57. Secondary Outcome: Change From Baseline Over Time in the Haemo-QoL-SF Questionnaire Physical Health Domain Score, as Completed by Treated Participants ≥8 to <12 Years of Age
Description: The Haemo-QoL-SF is a self-reported questionnaire for children ≥8 years of age. It contains 35 items, which cover nine domains considered relevant for the children's health-related quality of life: Physical Health, Feelings, View of Yourself, Family, Friends, Other People, Sports and School, Dealing with Hemophilia, and Treatment. The Physical Health domain assesses hemophilia-related symptoms (painful swellings and presence of joint pain) and physical functioning (pain with movement). Items are rated with five respective response options: never, seldom, sometimes, often, and always. The Physical Health domain score ranges from 0 to 100, with a lower score reflective of better physical health.
Time Frame: as for outcome 56
Population: as for outcome 56
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 22 | 6 | 6
units on a scale
  Baseline (value at visit): number analyzed (Participants) | 18 | 6 | 6
  Baseline (value at visit) | 29.51 [16.38 to 42.65] | 30.21 [21.49 to 38.93] | 19.79 [-7.23 to 46.81]
  Change from Baseline at Week 13: number analyzed (Participants) | 18 | 6 | 5
  Change from Baseline at Week 13 | -18.40 [-31.08 to -5.72] | -23.96 [-28.90 to -19.02] | 3.75 [-46.12 to 53.62]
  Change from Baseline at Week 25: number analyzed (Participants) | 18 | 6 | 4
  Change from Baseline at Week 25 | -18.40 [-33.76 to -3.05] | -17.71 [-26.43 to -8.99] | -17.19 [-61.94 to 27.57]
  Change from Baseline at Week 37: number analyzed (Participants) | 17 | 6 | 3
  Change from Baseline at Week 37 | -21.32 [-36.61 to -6.04] | -25.00 [-33.30 to -16.70] | -22.92 [-85.66 to 39.83]
  Change from Baseline at Week 49: number analyzed (Participants) | 17 | 5 | 3
  Change from Baseline at Week 49 | -15.44 [-25.74 to -5.15] | -23.75 [-40.57 to -6.93] | -25.00 [-96.15 to 46.15]
  Change from Baseline at Week 57: number analyzed (Participants) | 12 | 4 | 2
  Change from Baseline at Week 57 | -17.19 [-29.99 to -4.39] | -23.44 [-32.96 to -13.92] | -25.00 [-342.66 to 292.66]
  Change from Baseline at Week 81: number analyzed (Participants) | 12 | 3 | 0
  Change from Baseline at Week 81 | -14.06 [-26.97 to -1.15] | -16.67 [-25.63 to -7.70] |
  Change from Baseline at Week 105: number analyzed (Participants) | 9 | 3 | 0
  Change from Baseline at Week 105 | -16.67 [-45.29 to 11.96] | -20.83 [-29.80 to -11.87] |
  Change from Baseline at Week 129: number analyzed (Participants) | 7 | 0 | 0
  Change from Baseline at Week 129 | -12.50 [-45.71 to 20.71] |  |
  Change from Baseline at Week 153: number analyzed (Participants) | 4 | 0 | 0
  Change from Baseline at Week 153 | -21.88 [-66.72 to 22.97] |  |
  Change from Baseline at Week 177: number analyzed (Participants) | 2 | 0 | 0
  Change from Baseline at Week 177 | 6.25 [-152.58 to 165.08] |  |
  Change from Baseline at SC or ED: number analyzed (Participants) | 11 | 3 | 2
  Change from Baseline at SC or ED | -23.30 [-43.35 to -3.24] | -29.17 [-52.88 to -5.45] | -40.63 [-318.57 to 237.32]

58. Secondary Outcome: Change From Baseline Over Time in Caregiver-Reported Adapted Health-Related Quality of Life for Hemophilia Patients With Inhibitors Including Aspects of Caregiver Burden (Adapted Inhib-QoL) Questionnaire Total Score, Treated Participants <12 Years of Age
Description: Proxy assessment of health-related quality of life (HRQoL) and aspects of caregiver burden were assessed using the Adapted Inhib-QoL questionnaire, which comprises two parts with a total of 30 questions. The first part asks the caregiver for his/her opinion on the child's HRQoL and consists of two scales: Physical Health and Treatment. The second part asks the caregiver to rate how the child's situation is for them (i.e., the impact of the child's disease and treatment on the caregiver) and consists of 6 scales (5 if the child does not have siblings): General Condition, Dealing with the Inhibitor, Perceive Treatment, Family life, Siblings, Contact with Others. Items are rated with five respective response options: never, seldom, sometimes, often, and all the time. The Total Score is derived from the individual scores of all of the domains and it ranges from 0 to 100, with lower scores reflective of better HRQoL.
Time Frame: as for outcome 56
Population: All treated participants <12 years of age, as completed by their caregivers; at each timepoint, the number analyzed is the number of participants who completed a sufficient number of questionnaire items.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 65 | 10 | 10
units on a scale
  Baseline (value at visit): number analyzed (Participants) | 58 | 10 | 10
  Baseline (value at visit) | 43.10 [39.63 to 46.56] | 40.56 [32.46 to 48.65] | 31.45 [19.93 to 42.97]
  Change from Baseline at Week 13: number analyzed (Participants) | 58 | 10 | 9
  Change from Baseline at Week 13 | -19.76 [-23.55 to -15.96] | -21.46 [-27.21 to -15.72] | -9.24 [-21.69 to 3.21]
  Change from Baseline at Week 25: number analyzed (Participants) | 58 | 10 | 8
  Change from Baseline at Week 25 | -21.67 [-25.39 to -17.94] | -26.11 [-32.64 to -19.58] | -13.93 [-24.21 to -3.64]
  Change from Baseline at Week 37: number analyzed (Participants) | 57 | 10 | 7
  Change from Baseline at Week 37 | -21.79 [-25.30 to -18.28] | -24.62 [-32.28 to -16.97] | -12.55 [-25.73 to 0.64]
  Change from Baseline at Week 49: number analyzed (Participants) | 56 | 9 | 7
  Change from Baseline at Week 49 | -22.12 [-25.50 to -18.74] | -24.57 [-32.66 to -16.49] | -18.18 [-31.98 to -4.38]
  Change from Baseline at Week 57: number analyzed (Participants) | 41 | 7 | 6
  Change from Baseline at Week 57 | -20.86 [-24.87 to -16.85] | -24.37 [-34.52 to -14.22] | -20.28 [-39.65 to -0.92]
  Change from Baseline at Week 81: number analyzed (Participants) | 32 | 4 | 4
  Change from Baseline at Week 81 | -22.29 [-27.58 to -17.00] | -24.95 [-35.71 to -14.18] | -14.84 [-33.45 to 3.76]
  Change from Baseline at Week 105: number analyzed (Participants) | 20 | 4 | 4
  Change from Baseline at Week 105 | -18.04 [-26.73 to -9.34] | -21.82 [-43.00 to -0.64] | -15.82 [-31.09 to -0.55]
  Change from Baseline at Week 129: number analyzed (Participants) | 16 | 0 | 0
  Change from Baseline at Week 129 | -15.43 [-24.41 to -6.46] |  |
  Change from Baseline at Week 153: number analyzed (Participants) | 7 | 0 | 0
  Change from Baseline at Week 153 | -11.68 [-29.51 to 6.14] |  |
  Change from Baseline at Week 177: number analyzed (Participants) | 6 | 0 | 0
  Change from Baseline at Week 177 | -22.41 [-42.41 to -2.40] |  |
  Change from Baseline at SC or ED: number analyzed (Participants) | 52 | 6 | 4
  Change from Baseline at SC or ED | -23.59 [-27.38 to -19.80] | -25.83 [-36.77 to -14.89] | -13.73 [-52.15 to 24.69]

59. Secondary Outcome: Change From Baseline Over Time in the Caregiver-Reported Adapted Inhib-QoL Questionnaire Physical Health Domain Score, Treated Participants <12 Years of Age
Description: Proxy assessment of health-related quality of life (HRQoL) and aspects of caregiver burden were assessed using the Adapted Inhib-QoL questionnaire, which comprises two parts with a total of 30 questions. The first part asks the caregiver for his/her opinion on the child's HRQoL (proxy HRQoL) and consists of two scales: Physical Health and Treatment. The second part asks the caregiver to rate how the child's situation is for them (i.e., the impact of the child's disease and treatment on the caregiver) and consists of 6 scales (5 if the child does not have siblings): General Condition, Dealing with the Inhibitor, Perceive Treatment, Family Life, Siblings, Contact with Others. Items are rated with five respective response options: never, seldom, sometimes, often, and all the time. A total score is calculated as the sum of all of the items in the scale. The Physical Health domain score ranges from 0 to 100, with lower scores reflective of better physical health.
Time Frame: as for outcome 56
Population: as for outcome 58
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 65 | 10 | 10
units on a scale
  Baseline (value at visit): number analyzed (Participants) | 58 | 10 | 10
  Baseline (value at visit) | 37.13 [31.69 to 42.57] | 34.64 [18.13 to 51.16] | 20.00 [2.41 to 37.59]
  Change from Baseline at Week 13: number analyzed (Participants) | 58 | 10 | 9
  Change from Baseline at Week 13 | -31.10 [-36.78 to -25.42] | -30.00 [-46.83 to -13.17] | -6.35 [-33.24 to 20.54]
  Change from Baseline at Week 25: number analyzed (Participants) | 58 | 10 | 8
  Change from Baseline at Week 25 | -30.73 [-35.88 to -25.58] | -29.64 [-46.03 to -13.26] | -17.86 [-37.85 to 2.14]
  Change from Baseline at Week 37: number analyzed (Participants) | 57 | 10 | 7
  Change from Baseline at Week 37 | -31.20 [-36.66 to -25.75] | -31.07 [-46.45 to -15.69] | -21.94 [-43.97 to 0.09]
  Change from Baseline at Week 49: number analyzed (Participants) | 56 | 9 | 7
  Change from Baseline at Week 49 | -28.76 [-34.33 to -23.20] | -29.37 [-45.94 to -12.79] | -22.96 [-45.75 to -0.17]
  Change from Baseline at Week 57: number analyzed (Participants) | 41 | 7 | 6
  Change from Baseline at Week 57 | -27.79 [-33.94 to -21.63] | -32.65 [-50.38 to -14.92] | -26.19 [-54.20 to 1.82]
  Change from Baseline at Week 81: number analyzed (Participants) | 32 | 4 | 4
  Change from Baseline at Week 81 | -31.36 [-39.13 to -23.59] | -23.21 [-51.25 to 4.82] | -13.39 [-49.74 to 22.96]
  Change from Baseline at Week 105: number analyzed (Participants) | 20 | 4 | 4
  Change from Baseline at Week 105 | -27.86 [-40.08 to -15.64] | -18.75 [-59.83 to 22.33] | -16.96 [-44.17 to 10.24]
  Change from Baseline at Week 129: number analyzed (Participants) | 16 | 0 | 0
  Change from Baseline at Week 129 | -27.01 [-41.30 to -12.72] |  |
  Change from Baseline at Week 153: number analyzed (Participants) | 7 | 0 | 0
  Change from Baseline at Week 153 | -30.10 [-45.58 to -14.63] |  |
  Change from Baseline at Week 177: number analyzed (Participants) | 6 | 0 | 0
  Change from Baseline at Week 177 | -32.14 [-61.17 to -3.11] |  |
  Change from Baseline at SC or ED: number analyzed (Participants) | 52 | 6 | 4
  Change from Baseline at SC or ED | -30.29 [-36.26 to -24.32] | -35.12 [-58.99 to -11.25] | -21.43 [-79.38 to 36.53]

60. Secondary Outcome: Number of Participants With at Least One Adverse Event
Description: The number of participants experiencing at least one adverse event, including all non-serious and serious adverse events, are reported.
Time Frame: From Baseline up to 24 weeks after study drug discontinuation; the median (min-max) observation periods in Cohorts A, B, and C were 96.93 (36.1-188.1) weeks, 68.21 (56.7-129.4) weeks, and 69.43 (38.9-144.3) weeks, respectively.
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants | 64 | 9 | 10

61. Secondary Outcome: Number of Participants With at Least One Grade ≥3 Adverse Event
Description: The World Health Organization (WHO) toxicity grading scale was used for assessing adverse event severity. For adverse events that are not specifically listed in the WHO toxicity grading scale, a grade 3 adverse event is defined as: severe, marked limitation in activity, some assistance usually required, medical intervention or therapy required, hospitalization possible; and a grade 4 adverse event is defined as: life-threatening, extreme limitation in activity, significant assistance required, significant medical intervention or therapy required, hospitalization or hospice care probable.
Time Frame: as for outcome 60
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants | 15 | 1 | 3

62. Secondary Outcome: Number of Participants With at Least One Adverse Event Leading to Withdrawal From Treatment
Time Frame: as for outcome 60
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants | 0 | 0 | 1

63. Secondary Outcome: Number of Participants With at Least One Adverse Event of Local Injection Site Reaction
Description: Local adverse events that occurred within 24 hours after study drug administration and, in the investigator's opinion, were judged to be related to study drug injection, were captured as an "injection-site reaction" on the Adverse Event electronic Case Report Form (eCRF). An injection-related reaction that was localized was marked as a "local injection-site reaction."
Time Frame: as for outcome 60
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants | 23 | 2 | 6

64. Secondary Outcome: Number of Participants With at Least One Adverse Event of Systemic Hypersensitivity, Anaphylaxis, or Anaphylactoid Reaction
Description: Systemic hypersensitivity, anaphylaxis, or anaphylactoid reactions were identified by the investigator using Sampson's criteria, as defined in the protocol. At the primary completion date, one participant had reported two non-serious adverse events (cough and abdominal pain) that were identified as a potential case based on a Standardised MedDRA Queries (SMQ) search for Sampson's criteria. However, after medical review of the case, it was confirmed that this case was not indicative of a systemic hypersensitivity, anaphylaxis, or anaphylactoid reaction.
Time Frame: as for outcome 60
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants | 1 | 0 | 0

65. Secondary Outcome: Number of Participants With at Least One Adverse Event of Thromboembolic Event
Time Frame: as for outcome 60
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants | 0 | 0 | 0

66. Secondary Outcome: Number of Participants With at Least One Adverse Event of Thrombotic Microangiopathy
Time Frame: as for outcome 60
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants | 0 | 0 | 0

67. Secondary Outcome: Number of Participants Testing Negative or Positive for the Presence of Anti-Drug Antibodies (ADAs), Including Neutralizing ADAs, During the Study
Description: 'Total ADA Negative' is the sum of all subjects who tested negative for ADA in the 2 following categories: 'ADA Negative', those who are pre-dose ADA negative or are missing pre-dose ADA data and who have all negative post-dose ADA results; and 'ADA Negative (Treatment Unaffected)', a subset who are pre-dose ADA positive but do not have a ≥4-fold increase in post-dose ADA levels compared to baseline measurement. 'Total ADA Positive' is the sum of all subjects who tested positive for ADA in the 2 following categories: 'ADA Positive (Treatment Boosted)', those who are pre-dose ADA positive and have a ≥4-fold increase in post-dose ADA levels compared to baseline measurement; and 'ADA Positive (Treatment Induced)', those who are pre-dose ADA negative or missing data and who have at least one post-dose ADA positive sample. ADA-positive samples were further analyzed for neutralizing capacity using a modified FVIII chromogenic assay; if also positive, they were considered neutralizing ADAs.
Time Frame: Predose (0 hour) at Weeks 1, 5, 17, 33, 49, 57; then every 12 weeks until study completion (up to 188 weeks)
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants
  Total ADA Negative (Neg + Neg Unaffected) | 63 | 10 | 9
  ADA Negative | 59 | 10 | 9
  ADA Negative (Treatment Unaffected) | 4 | 0 | 0
  Total ADA Positive (Boosted + Induced) | 5 | 0 | 1
  ADA Positive (Treatment Boosted) | 0 | 0 | 0
  ADA Positive (Treatment Induced) | 5 | 0 | 1
  ADA Positive with Neutralizing ADAs | 2 | 0 | 1

68. Secondary Outcome: Number of Participants by Hematology Parameter Laboratory Test Results as a Shift From Baseline to Highest WHO Grade Post-Baseline
Description: The World Health Organization (WHO) toxicity grading scale was used for determining the severity of laboratory abnormalities (i.e., test results outside of the reference range) for hematology parameters; Grade 0 is normal and Grades 1 to 4 represent worsening levels of the parameter outside of the normal range in the specified direction of the abnormality (high and low are above and below the range, respectively). Not every laboratory abnormality qualified as an adverse event (AE). A laboratory test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment. Baseline was defined as the last available assessment prior to first receipt of study drug. Abs = absolute count
Time Frame: From Baseline until study completion (up to 188 weeks)
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants
  Hemoglobin, Low - Grade 0 to 0 | 53 | 10 | 9
  Hemoglobin, Low - Grade 0 to 1 | 3 | 0 | 1
  Hemoglobin, Low - Grade 0 to 2 | 4 | 0 | 0
  Hemoglobin, Low - Grade 1 to 0 | 3 | 0 | 0
  Hemoglobin, Low - Grade 1 to 1 | 4 | 0 | 0
  Hemoglobin, Low - Grade 2 to 2 | 1 | 0 | 0
  Neutrophils (Total, Abs), Low - Grade 0 to 0 | 39 | 7 | 9
  Neutrophils (Total, Abs), Low - Grade 0 to 1 | 14 | 1 | 1
  Neutrophils (Total, Abs), Low - Grade 0 to 2 | 5 | 2 | 0
  Neutrophils (Total, Abs), Low - Grade 0 to 3 | 3 | 0 | 0
  Neutrophils (Total, Abs), Low - Grade 0 to 4 | 1 | 0 | 0
  Neutrophils (Total, Abs), Low - Grade 1 to 1 | 4 | 0 | 0
  Neutrophils (Total, Abs), Low - Grade 1 to 2 | 1 | 0 | 0
  Neutrophils (Total, Abs), Low - Grade 1 to 3 | 1 | 0 | 0
  Platelets, Low - Grade 0 to 0 | 68 | 8 | 10
  Platelets, Low - Grade 0 to 1 | 0 | 2 | 0

69. Secondary Outcome: Number of Participants by Chemistry Parameter Laboratory Test Results as a Shift From Baseline to Highest WHO Grade Post-Baseline
Description: The World Health Organization (WHO) toxicity grading scale was used for determining the severity of laboratory abnormalities (i.e., test results outside of the reference range) for chemistry parameters; Grade 0 is normal and Grades 1 to 4 represent worsening levels of the parameter outside of the normal range in the specified direction of the abnormality (high and low are above and below the range, respectively). Not every laboratory abnormality qualified as an adverse event (AE). A laboratory test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment. Baseline was defined as the last available assessment prior to first receipt of study drug. SGOT/AST = aspartate aminotransferase; SGPT/ALT = alanine aminotransferase
Time Frame: From Baseline until study completion (up to 188 weeks)
Population: All participants who received at least one dose of emicizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
Participants
  Alkaline Phosphatase, High - Grade 0 to 0 | 49 | 8 | 6
  Alkaline Phosphatase, High - Grade 0 to 1 | 4 | 1 | 0
  Alkaline Phosphatase, High - Grade 0 to 2 | 2 | 0 | 0
  Alkaline Phosphatase, High - Grade 1 to 1 | 6 | 1 | 2
  Alkaline Phosphatase, High - Grade 1 to 2 | 3 | 0 | 1
  Alkaline Phosphatase, High - Grade 2 to 1 | 1 | 0 | 0
  Alkaline Phosphatase, High - Grade 2 to 2 | 1 | 0 | 0
  Alkaline Phosphatase, High - Missing to Grade 0 | 0 | 0 | 1
  Alkaline Phosphatase, High - Missing to Grade 3 | 2 | 0 | 0
  Bilirubin, High - Grade 0 to 0 | 62 | 10 | 10
  Bilirubin, High - Grade 0 to 1 | 1 | 0 | 0
  Bilirubin, High - Grade 0 to 2 | 2 | 0 | 0
  Bilirubin, High - Missing to Grade 0 | 3 | 0 | 0
  Blood Urea Nitrogen, High - Grade 0 to 0 | 58 | 10 | 9
  Blood Urea Nitrogen, High - Grade 0 to 1 | 3 | 0 | 1
  Blood Urea Nitrogen, High - Grade 1 to 1 | 3 | 0 | 0
  Blood Urea Nitrogen, High - Missing to Grade 0 | 1 | 0 | 0
  Blood Urea Nitrogen, High - Missing to Grade 1 | 1 | 0 | 0
  Blood Urea Nitrogen, High - Missing to Grade 2 | 2 | 0 | 0
  Calcium (Corrected), Low - Grade 0 to 0 | 54 | 7 | 9
  Calcium (Corrected), Low - Grade 0 to 1 | 5 | 3 | 0
  Calcium (Corrected), Low - Grade 0 to 2 | 2 | 0 | 0
  Calcium (Corrected), Low - Grade 0 to 4 | 1 | 0 | 0
  Calcium (Corrected), Low - Missing to Grade 0 | 5 | 0 | 1
  Calcium (Corrected), Low - Missing to Grade 2 | 1 | 0 | 0
  Calcium (Corrected), High - Grade 0 to 0 | 61 | 10 | 9
  Calcium (Corrected), High - Grade 2 to 0 | 1 | 0 | 0
  Calcium (Corrected), High - Missing to Grade 0 | 6 | 0 | 1
  Creatinine, High - Grade 0 to 0 | 62 | 9 | 9
  Creatinine, High - Grade 0 to 1 | 5 | 1 | 0
  Creatinine, High - Grade 1 to 1 | 1 | 0 | 1
  Glucose, Low - Grade 0 to 0 | 57 | 8 | 8
  Glucose, Low - Grade 0 to 1 | 6 | 2 | 1
  Glucose, Low - Grade 0 to 2 | 1 | 0 | 0
  Glucose, Low - Grade 0 to 3 | 1 | 0 | 0
  Glucose, Low - Grade 1 to 0 | 0 | 0 | 1
  Glucose, Low - Grade 2 to 0 | 1 | 0 | 0
  Glucose, Low - Missing to Grade 0 | 1 | 0 | 0
  Glucose, Low - Missing to Grade 1 | 1 | 0 | 0
  Glucose, High - Grade 0 to 0 | 31 | 5 | 4
  Glucose, High - Grade 0 to 1 | 28 | 3 | 6
  Glucose, High - Grade 0 to 2 | 4 | 0 | 0
  Glucose, High - Grade 1 to 0 | 1 | 1 | 0
  Glucose, High - Grade 1 to 1 | 1 | 0 | 0
  Glucose, High - Grade 2 to 1 | 1 | 0 | 0
  Glucose, High - Grade 2 to 3 | 0 | 1 | 0
  Glucose, High - Missing to Grade 0 | 1 | 0 | 0
  Glucose, High - Missing to Grade 1 | 1 | 0 | 0
  Magnesium, Low - Grade 0 to 0 | 57 | 9 | 9
  Magnesium, Low - Grade 0 to 1 | 6 | 1 | 1
  Magnesium, Low - Grade 4 to 1 | 1 | 0 | 0
  Magnesium, Low - Missing to Grade 0 | 3 | 0 | 0
  Magnesium, Low - Missing to Grade 2 | 1 | 0 | 0
  Phosphorus, Low - Grade 0 to 0 | 64 | 10 | 10
  Phosphorus, Low - Missing to Grade 0 | 4 | 0 | 0
  Potassium, Low - Grade 0 to 0 | 61 | 9 | 10
  Potassium, Low - Grade 0 to 1 | 5 | 1 | 0
  Potassium, Low - Grade 0 to 2 | 1 | 0 | 0
  Potassium, Low - Grade 1 to 0 | 1 | 0 | 0
  Potassium, High - Grade 0 to 0 | 66 | 10 | 10
  Potassium, High - Grade 0 to 1 | 1 | 0 | 0
  Potassium, High - Grade 0 to 4 | 1 | 0 | 0
  SGOT/AST, High - Grade 0 to 0 | 54 | 8 | 9
  SGOT/AST, High - Grade 0 to 1 | 9 | 1 | 1
  SGOT/AST, High - Grade 0 to 2 | 1 | 0 | 0
  SGOT/AST, High - Grade 1 to 1 | 3 | 0 | 0
  SGOT/AST, High - Missing to Grade 1 | 1 | 1 | 0
  SGPT/ALT, High - Grade 0 to 0 | 52 | 10 | 9
  SGPT/ALT, High - Grade 0 to 1 | 8 | 0 | 0
  SGPT/ALT, High - Grade 0 to 2 | 4 | 0 | 0
  SGPT/ALT, High - Grade 0 to 3 | 1 | 0 | 0
  SGPT/ALT, High - Grade 1 to 1 | 2 | 0 | 1
  SGPT/ALT, High - Missing to Grade 0 | 1 | 0 | 0
  Sodium, Low - Grade 0 to 0 | 45 | 8 | 8
  Sodium, Low - Grade 0 to 1 | 18 | 1 | 0
  Sodium, Low - Grade 0 to 2 | 2 | 0 | 0
  Sodium, Low - Grade 1 to 0 | 0 | 0 | 2
  Sodium, Low - Grade 1 to 1 | 2 | 1 | 0
  Sodium, Low - Grade 1 to 2 | 1 | 0 | 0
  Sodium, High - Grade 0 to 0 | 58 | 9 | 10
  Sodium, High - Grade 0 to 1 | 8 | 1 | 0
  Sodium, High - Grade 0 to 2 | 1 | 0 | 0
  Sodium, High - Grade 0 to 4 | 1 | 0 | 0

70. Secondary Outcome: Plasma Trough Concentration (Ctrough) of Emicizumab
Description: Pre-dose (trough) plasma concentrations of emicizumab were analyzed using a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantitation was 0.1 micrograms per milliliter (μg/mL).
Time Frame: Predose (0 hour) at Weeks 1, 2, 3, 4, 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 49, 57, 69, 81, 93, 105, 117, 129, 141, 153, 165, and 177
Population: Participants who received at least one dose of emicizumab and had at least one post-dose emicizumab plasma concentration result available
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
Number analyzed (Participants) | 68 | 10 | 10
micrograms per milliliter (μg/mL)
  Week 1: number analyzed (Participants) | 67 | 10 | 10
  Week 1 | NA (NA) — No data available because the measurements were below the limit of quantitation. | NA (NA) — No data available because the measurements were below the limit of quantitation. | NA (NA) — No data available because the measurements were below the limit of quantitation.
  Week 2: number analyzed (Participants) | 66 | 10 | 10
  Week 2 | 18.2 (5.5) | 17.0 (3.9) | 17.2 (4.1)
  Week 3: number analyzed (Participants) | 67 | 10 | 9
  Week 3 | 31.6 (5.6) | 31.7 (6.8) | 33.9 (5.8)
  Week 4: number analyzed (Participants) | 67 | 10 | 10
  Week 4 | 42.9 (8.0) | 42.4 (9.5) | 44.7 (7.0)
  Week 5: number analyzed (Participants) | 66 | 10 | 9
  Week 5 | 53.3 (10.6) | 51.8 (10.5) | 56.4 (12.3)
  Week 7: number analyzed (Participants) | 68 | 10 | 8
  Week 7 | 51.2 (10.5) | 51.5 (9.6) | 59.9 (24.6)
  Week 9: number analyzed (Participants) | 67 | 10 | 9
  Week 9 | 49.9 (9.7) | 51.9 (11.2) | 39.3 (16.7)
  Week 13: number analyzed (Participants) | 67 | 10 | 9
  Week 13 | 48.3 (13.3) | 45.3 (10.8) | 37.1 (10.6)
  Week 17: number analyzed (Participants) | 68 | 10 | 8
  Week 17 | 46.1 (11.2) | 48.7 (10.4) | 36.3 (6.1)
  Week 21: number analyzed (Participants) | 67 | 10 | 8
  Week 21 | 45.2 (11.1) | 43.9 (11.0) | 36.2 (12.4)
  Week 25: number analyzed (Participants) | 68 | 10 | 8
  Week 25 | 46.9 (11.7) | 41.9 (8.5) | 33.7 (8.9)
  Week 29: number analyzed (Participants) | 68 | 9 | 8
  Week 29 | 47.9 (13.0) | 46.7 (5.1) | 34.4 (9.0)
  Week 33: number analyzed (Participants) | 67 | 10 | 7
  Week 33 | 51.3 (13.8) | 51.0 (6.8) | 34.7 (11.2)
  Week 37: number analyzed (Participants) | 66 | 9 | 7
  Week 37 | 51.0 (15.3) | 50.4 (6.4) | 35.9 (9.1)
  Week 41: number analyzed (Participants) | 66 | 10 | 7
  Week 41 | 48.5 (14.2) | 55.3 (10.7) | 38.1 (9.9)
  Week 49: number analyzed (Participants) | 66 | 10 | 7
  Week 49 | 49.4 (12.6) | 48.6 (9.2) | 32.4 (7.5)
  Week 57: number analyzed (Participants) | 60 | 9 | 6
  Week 57 | 46.2 (15.9) | 46.4 (9.8) | 28.5 (10.7)
  Week 69: number analyzed (Participants) | 52 | 4 | 4
  Week 69 | 46.4 (16.0) | 54.7 (11.5) | 41.1 (5.2)
  Week 81: number analyzed (Participants) | 36 | 4 | 4
  Week 81 | 45.6 (14.2) | 38.0 (5.3) | 35.7 (21.2)
  Week 93: number analyzed (Participants) | 34 | 4 | 4
  Week 93 | 44.3 (13.8) | 41.2 (6.6) | 41.6 (26.8)
  Week 105: number analyzed (Participants) | 22 | 4 | 4
  Week 105 | 46.9 (15.9) | 43.4 (5.7) | 34.2 (14.4)
  Week 117: number analyzed (Participants) | 19 | 4 | 4
  Week 117 | 37.8 (12.3) | 46.6 (10.2) | 37.1 (12.9)
  Week 129: number analyzed (Participants) | 18 | 0 | 0
  Week 129 | 39.7 (13.8) |  |
  Week 141: number analyzed (Participants) | 17 | 0 | 0
  Week 141 | 46.5 (17.2) |  |
  Week 153: number analyzed (Participants) | 12 | 0 | 0
  Week 153 | 39.5 (15.6) |  |
  Week 165: number analyzed (Participants) | 11 | 0 | 0
  Week 165 | 39.9 (17.8) |  |
  Week 177: number analyzed (Participants) | 12 | 0 | 0
  Week 177 | 38.9 (19.0) |  |

ADVERSE EVENTS:
Time Frame: From Baseline up to 24 weeks after study drug discontinuation; the median (min-max) observation periods in Cohorts A, B, and C were 96.93 (36.1-188.1) weeks, 68.21 (56.7-129.4) weeks, and 69.43 (38.9-144.3) weeks, respectively.
Arm/Group | Cohort A: 1.5 mg/kg Emicizumab QW | Cohort B: 3 mg/kg Emicizumab Q2W | Cohort C: 6 mg/kg Emicizumab Q4W
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 23/68 | 1/10 | 3/10
Other Adverse Events (participants affected / at risk) | 64/68 | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: 1.5 mg/kg Emicizumab QW (N=68) | Cohort B: 3 mg/kg Emicizumab Q2W (N=10) | Cohort C: 6 mg/kg Emicizumab Q4W (N=10)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Neutralising antibodies positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: 1.5 mg/kg Emicizumab QW (N=68) | Cohort B: 3 mg/kg Emicizumab Q2W (N=10) | Cohort C: 6 mg/kg Emicizumab Q4W (N=10)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 12 (16) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (15) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 22 (44) | 2 (6) | 6 (19)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 21 (44) | 6 (8) | 4 (5)
Swelling face (General disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 7 (10) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (7) | 0 (0) | 1 (2)
Ear infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (9) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 8 (13) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 29 (53) | 3 (11) | 4 (10)
Otitis media (Infections and infestations) | 7 (8) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (4) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (2)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsilitis (Infections and infestations) | 7 (13) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 23 (44) | 0 (0) | 2 (2)
Varicella (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 11 (70) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 10 (21) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 5 (6) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (11) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 6 (6) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 8 (15) | 0 (0) | 0 (0)
Indeterminable ABO blood type (Investigations) | 1 (1) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (19) | 2 (2) | 2 (13)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 3 (5)
Headache (Nervous system disorders) | 12 (17) | 1 (10) | 2 (2)
Device breakage (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (28) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 2 (4) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 5 (7) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 1 (1)
Vaccination site erythema (General disorders) | 3 (3) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 4 (4) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 4 (7) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02795767/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02795767/SAP_001.pdf